CLINICAL TRIAL: NCT03209297
Title: The Effect of Conservative Treatment of Temporomandibular Disorders on Somatic Tinnitus
Brief Title: Temporomandibular Dysfunction in Patients With Tinnitus: Assessment and Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Collaborators: University Hospital, Antwerp (Other); Fonds voor Wetenschappelijk onderzoek Vlaanderen (Unknown)
Responsible Party: Principal Investigator, Sarah Michiels, Post-doctoral researcher, Universiteit Antwerpen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: T001916N
Record Dates: First submitted 2017-04-19; First posted 2017-07-06 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Tinnitus, Subjective
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Intervention Model Description: One study arm will be treated immediately after inclusion. The other study arm will be treated after a delay of 9 weeks. During these 9 weeks patients will be on a waiting list.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Direct treatment (Experimental): Patients receive the TMD treatment immediately
  Interventions: Other: TMD treatment: physiotherapy and/or occlusal splints
- Delayed treatment (Experimental): No intervention in the first 9 weeks of the study. Afterwards, the patients receive the same treatment as the other group
  Interventions: Other: TMD treatment: physiotherapy and/or occlusal splints

INTERVENTIONS:
Other: TMD treatment: physiotherapy and/or occlusal splints — The patient will receive the most appropriate TMD treatment, based on current literature.

SUMMARY:
TMD treatment, based on state of the art knowledge derived from clinical studies will be applied in patients with tinnitus and TMD. When this approach proves to be useful for the treatment of tinnitus, it offers a new therapeutic option for patients with tinnitus. To understand how TMD treatment works for patients with tinnitus, we will analyse mediating factors, i.e. factors that contribute to the therapeutic effect. To help clinicians in their clinical process we will identify prognostic indicators, i.e. factors that predict a positive or negative outcome of TMD treatment. This can provide a helpful tool in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included when suffering from somatic tinnitus, attributed to TMD, which has been stable for at least 3 months.
* Tinnitus Functional Index score between 25 and 90

Exclusion Criteria:

* clear otological or neurological causes of the tinnitus such as Menière's disease, severe depression (diagnosed by a psychologist), progressive middle ear pathology, intracranial pathology
* traumatic cervical spine or temporomandibular injury in the past 6 months
* tumours
* previous surgery in the orofacial area
* in case physical therapy treatment directed to the orofacial area is contra-indicated
* if the patient received TMD treatment in the past 2 months
* drug intake that can affect the outcome measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-11-05 (Actual)

PRIMARY OUTCOMES:
Tinnitus Questionnaire | Baseline, 9 weeks, 18 weeks, 27 weeks
  Questionnaire to measure the change in tinnitus related distress

SECONDARY OUTCOMES:
Tinnitus Functional Index | Baseline, 9 weeks, 18 weeks, 27 weeks
  Questionnaire to measure the change in tinnitus severity
Hyperacusis Questionnaire | Baseline
  Questionnaire to measure the presence of hyperacusis
Visual analogue scale for tinnitus loudness | Baseline, 9 weeks, 18 weeks, 27 weeks
  Scale to measure the change in average tinnitus loudness
TMD pain screener | Baseline, 9 weeks, 18 weeks, 27 weeks
  Questionnaire to assess the presence of and change in temporomandibular disorders(TMD) symptoms
Hospital anxiety and depression scale | Baseline
  Questionnaire to measure the presence of anxiety and/or depression
Specific anamnestic questions | Baseline
  pre-defined list of questions on duration of the tinnitus complaints, modulation, bruxism,...
Static investigation of the temporomandibular joint | Baseline, 9 weeks, 18 weeks, 27 weeks
  evaluation of change in isometric contraction of jaw muscles
Dynamic investigation of the temporomandibular joint | Baseline, 9 weeks, 18 weeks, 27 weeks
  evaluation of change in isotonic contraction of jaw muscles
Pain pressure threshold | Baseline, 9 weeks, 18 weeks, 27 weeks
  measurement of change in pain pressure thresholds on masseter, temporalis, temporomandibular joint, sternocleidomastoideus, tibialis anterior
Mouth opening | Baseline, 9 weeks, 18 weeks, 27 weeks
  change in mouth opening measured in cm with a ruler
Pain on palpation of masseter, temporalis and temporomandibular joint | Baseline, 9 weeks, 18 weeks, 27 weeks
  change in recognisable pain on palpation, measured on numerical rating scale
Tinnitus Analysis | Baseline
  analysis of the tinnitus type, pitch and loudness
Speech in noise test | Baseline, 9 weeks, 18 weeks, 27 weeks
  analysis of the change in understanding spoken words in a noisy situation
Pure tone audiometry | Baseline
  evaluation of possible hearing problems
Auditory evoked potentials measurement | Baseline, 18 weeks
  change in EEG during listening tasks

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair ziekenhuis Antwerpen, Edegem, Antwerpen, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Michiels S, van der Wal AC, Nieste E, Van de Heyning P, Braem M, Visscher C, Topsakal V, Gilles A, Jacquemin L, Hesters M, De Hertogh W. Conservative therapy for the treatment of patients with somatic tinnitus attributed to temporomandibular dysfunction: study protocol of a randomised controlled trial. Trials. 2018 Oct 12;19(1):554. doi: 10.1186/s13063-018-2903-1. PMID 30314506